姓 名: 生 日:西元 年 月 日

# 國立臺灣大學醫學院附設醫院 National Taiwan University Hospital

# 臨床試驗/研究受試者說明暨同意書

研究倫理委員會案號: 202201057RINA

請詳細閱讀內容,待主持人或其授權人員向您說明後,再簽署同意書

第1頁

# 計書名稱

中文:標定巨噬細胞與癌細胞融合機制以改善癌症纖維增生

英文: Targeting fusion machinery between macrophages and cancer

cells to ameliorate cancer desmoplasia

試驗機構:台大醫院 內 科/部

委託單位/藥廠:無

研究經費來源:國衛院

試驗主持人:姚明

職稱:內科部 主治醫師 主任

協同主持人:羅仕錡

職稱:檢醫部 主治醫師 主任

常慧如

職稱:國衛院癌研所 主治醫師

聯絡人:常慧如

上班時間聯絡電話:0911200099

受試者姓名:

病歷號碼:

您被邀請參與此臨床研究,這份表格提供您本研究之相關資訊,試驗主持人或其授權人 員將會為您說明研究內容並回答您的任何疑問。

在您的問題尚未獲得滿意的答覆之前,請不要簽署此同意書。您不須立即決定是否參加 本研究,請您經過慎重考慮後方予簽名。

您須簽署同意書後才能參與本研究。如果您願意參與本研究,此文件將視為您的同意紀錄。即使在您同意後,您仍然可以隨時退出本研究而不需理由。

以下內容為試驗之詳細程序及您應知事項,仍請您務必詳細閱讀。

## (一)試驗/研究目的:

這是一個研究正常巨噬血球細胞,造成癌細胞組織纖維化的研究. 因為您有正常的周邊血液,因此被邀請加入這個研究.

#### (二)研究背景:

癌症纖維增生,尤其在胰臟癌,是導致癌症惡化,對治療產生抗藥性的主要原因之一. 目前針對剔除被癌症活化之纖維細胞的治療,效果不如預期,反而會導致更具侵略性的癌症, 吸引抑制免疫反應的淋巴細胞,大量湧入腫瘤微環境.

考量巨噬細胞在發炎反應,纖維化,癌症發生,與惡化的角色,許多針對巨噬細胞剔除或極化的治療發展,得到具有潛力的臨床前期結果.研究顯示巨噬細胞與癌細胞的細胞融合,是導致腫瘤多樣性的動力,引起抗藥性與癌症惡化.但對於巨噬細胞與癌細胞的細胞融合,

在癌症纖維增生的研究很少. 版本/日期: 20220225 version 2

NTUHREC\_Version: AF- 046/09.0

西元 2017年 06月 19日病歷委員會修正通過 MR19-304 西元 2017年 05月 31日品質暨病人安全委員會審核通過

文件編號 01010-4-601566

姓 名: 日:西元 年月日

# 國立臺灣大學醫學院附設醫院 National Taiwan University Hospital

# 臨床試驗/研究受試者說明暨同意書

研究倫理委員會案號: 202201057RINA

請詳細閱讀內容,待主持人或其授權人員向您說明後,再簽署同意書

為改善胰臟癌治療效果,提高醫療經費經濟效益與病患生活品質,我們將發展以巨噬細 胞為主的治療策略,改善癌症纖維化環境,達到預防腫瘤新生、惡化,以及提高治療效果的目 的.

我們預計納入30位具有正常周邊血液的受試者,收集血液中的單核白血球,將其分化 為巨噬細胞, 在實驗室中與癌細胞共培養或融合, 研究巨噬與癌細胞的交互作用, 以及融合細 胞產生的生物特性,與纖維化特徵.

本研究不涉及藥品或醫療技術/器材.

## (三)研究之納入與排除條件:

執行本研究計畫的醫師或相關研究人員將會與您討論有關參加本研究的必要條件。請您配合 必須誠實告知我們您過去的健康情形,若您有不符合參加本研究的情況,將不能參加本研究計畫。

- 1. 納入條件(參加本研究的條件):
  - (1) 於進案一周內,有正常的周邊血液檢測結果.
  - (2) 若為捐髓者,可以為接受血球刺激或生長激素之後.
  - (3) 可以為血紅素偏高的放血者.
  - (4) 年龄 20-70歲.
- 2. 排除條件(若您有下列任一情況,您將無法參加本研究):
  - (1)有惡性腫瘤,且無復發狀態少於五年者.
  - (2)有重大心血管疾病, 免疫疾病, 懷孕.
  - (3)長期服用免疫抑制劑或類固醇者.

#### (四)本研究方法及相關程序:

您同意加入本研究後, 將以針筒由手臂, 抽取周邊血液10-20 ml, 置於添加抗凝血劑的 試管中, 血液檢體將初步處理, 分離出單核白血球後, 運送並儲存到台大姚明醫師, 或國衛院 常慧如醫師實驗室, 安排後續實驗: 包括分化為巨噬細胞, 與癌細胞共培養或融合, 進行融合 與未融合癌細胞惡性度研究. 有極小可能您的血球與癌細胞之融合細胞, 會形成細胞株, 繁 **殖一段時間, 但無論細胞株或**您的剩餘血液將儲存不超過10年,

本研究計畫也將回溯收集曾經接受骨髓移植、又發生腫瘤的病患之腫瘤組織檢體、進行 癌細胞是否與捐髓者巨噬細胞融合而來的研究.

除了為篩選進案所需基本資料與周邊血液數據,我們不會收集您的其他臨床資料,

版本/日期: 20220225 version 2

NTUHREC Version: AF- 046/09.0

西元 2017 年 06 月 19 日病歷委員會修正通過 MR19-304 西元 2017年 05月 31日品質暨病人安全委員會審核通過

01010-4-601566 文件編號

姓 名:

日:西元

國立臺灣大學醫學院附設醫院 National Taiwan University Hospital

臨床試驗/研究受試者說明暨同意書

年 月 日 研究倫理委員會案號: 202201057RINA

請詳細閱讀內容,待主持人或其授權人員向您說明後,再簽署同意書

第3頁

## (五)可能發生之風險及其發生率與處理方法:

您加入本研究,接收抽血,可能發生抽血部位少量出血,紅腫瘀血.極少情況有量眩的 情形、您只需靜坐一段時間、按壓抽血傷口止血、局部適度冰敷即可、若仍不適、可以詢求 醫護協助.

### (六)其他替代療法及說明:

本研究本身不牽涉治療,您的病情經醫師診療後,可考慮的標準治療方式包括藥物治療 手術治療等。如果您對治療有任何疑問請進一步與您的醫師討論。您可以拒絕加入研究,避 免額外的抽血量.

#### (七)試驗/研究預期效益:

目前無法預測可能的研究成果。當您的檢體使用於研究時,我們將不會通知您研究結果 或檢體的檢測結果。一般而言,研究所做的檢測分析,大多還不能運用於醫療照護;但若研 究人員認為研究分析的結果,有助於您的醫療照護,也可能會通知您。

## (八)試驗/研究進行中受試者之禁忌、限制與應配合之事項:

請配合抽血,沒有禁忌.

#### (九)受試者個人資料之保密:

台大醫院將依法,把任何可辨識您的身分之記錄,與您的個人隱私資料視為機密來處 理,不會公開。研究人員將以一個研究代碼代表您的身分,此代碼不會顯示您的姓名、國民 身分證統一編號、住址等可識別資料。如果發表研究結果,您的身分仍將保密。您亦瞭解若 簽署同意書,即同意您的原始醫療紀錄可直接受監測者、稽核者、研究倫理委員會及主管機 關(若試驗受美國食品藥物管理局管轄,則主管機關包含美國食品藥物管理局)檢閱,以確保 臨床研究過程, 與數據符合相關法律及法規要求. 上述人員並承諾絕不違反您的身分之機密 性。除了上述機構依法有權檢視外,我們會小心維護您的隱私。

#### (十)研究之退出與中止:

您可自由決定是否參加本研究;研究過程中也可隨時撤銷或中止同意,退出研究,不需 任何理由,且不會引起任何不愉快或影響其日後醫師對您的醫療照顧。

當您退出本研究,或主持人判斷您不適合繼續參與本研究時,在退出前已得到的資料將 被保留,不會移除。在退出後,您可選擇如何處理您先前提供的檢體,與決定是否同意試驗

版本/日期: 20220225 version 2

NTUHREC Version: AF- 046/09.0

西元 2017 年 06 月 19 日病歷委員會修正通過 MR19-304 西元 2017年 05月 31日品質暨病人安全委員會審核通過

01010-4-601566 文件編號

國立臺灣大學醫學院附設醫院 National Taiwan University Hospital

# B: 西元 年月日 臨床試驗/研究受試者說明暨同意書

研究倫理委員會案號: 202201057RINA

請詳細閱讀內容,待主持人或其授權人員向您說明後,再簽署同意書

第4頁

| 主持人繼續收集您的資料。 | <b>丰</b> 你的資料。 | 隼 | 收 | 繼續 | 人 | 丰持 |
|--------------|----------------|---|---|----|---|----|
|--------------|----------------|---|---|----|---|----|

- 1. 對我先前所提供的檢體
- □我同意繼續授權本研究使用於本試驗疾病相關的研究。逾越原書面同意使用範圍時, 需再次經過我同意。
- □不同意繼續授權本研究使用,但為確保已完成檢查之準確性,同意研究相關檢體可由 實驗室進行再次確認後銷毀。
- □不同意繼續授權本研究使用,請自我退出日起銷毀我之前的本研究相關檢體。
- 2. 退出後讓試驗主持人繼續收集我的資料,例如經由我的病歷記載取得後續醫療過程、實驗室檢查結果。繼續收集資料期間,仍會維護您的隱私和個人資料的機密性。
- □同意收集。
- □不同意本研究繼續收集或檢視我的資料,但可經由公共資料庫查詢之紀錄不在此限。

# (十一) 損害補償與保險:

試驗/研究一定有風險,為確保因為參與研究發生不良反應致造成您的損害時所可能獲得 之保障,請您務必詳閱本項說明內容:

- 如依本研究所訂臨床研究計畫,因發生不良反應造成損害,由台灣大學醫學院附設醫院 負補償責任。但本受試者同意書上所記載之可預期不良反應,不予補償。
- 2. 如依本研究所訂臨床研究計畫,因而發生不良反應或損害,本醫院願意提供專業醫療照 顧及醫療諮詢。您不必負擔治療不良反應或損害之必要醫療費用。
- 3.除前二項補償及醫療照顧外,本研究不提供其他形式之補償。若您不願意接受這樣的風險,請勿參加研究。
- 4. 您不會因為簽署本同意書,而喪失在法律上的任何權利。
- 5. 本研究未投保人體試驗責任保險。

若您確因參與本研究因而發生不良反應造成之損害,前述補償包括合理的醫療費用,惟應符合以下條件:您的損害並非故意造成;您遵守試驗醫師之醫療建議。

# (十二)受試者之檢體(含其衍生物)、個人資料之保存、使用與再利用

- 1. 檢體及剩餘檢體之保存與使用
  - (1)檢體(含其衍生物)之保存與使用

為研究所需,我們所蒐集您的檢體,將依本研究計畫使用,檢體將保存於<u>台大醫院</u> 內科部姚明醫師實驗室 及 國家衛生研究院癌症研究所常慧如醫師實驗室,直至 <u>2032</u>

#### 版本/日期: 20220225 version 2

NTUHREC\_Version: AF- 046/09.0

西元 2017年 06月 19日病歷委員會修正通過 MR19-304 西元 2017年 05月 31日品質暨病人安全委員會審核通過

文件編號 01010-4-601566

日:西元

## 國立臺灣大學醫學院附設醫院 National Taiwan University Hospital

# 臨床試驗/研究受試者說明暨同意書

年 月 日 研究倫理委員會案號: 202201057RINA

請詳細閱讀內容,待主持人或其授權人員向您說明後,再簽署同意書

年保存期限屆滿,我們將依法銷毀。為了保護您的個人隱私,我們將以一個研究編號來 代替您的名字及相關個人資料,以確認您的檢體及與相關資料受到完整保密。如果您對 檢體的使用有疑慮,或您有任何想要銷毀檢體的需求,請立即與我們聯絡 (聯絡人:常 慧如電話: 0911200099 ; 聯絡單位: 國家衛生研究院癌症研究所 電話: 037-246166 ext 35105 地址: 苗栗縣竹南鎮科研路 35 號 R1-2034 室), 我們即會將您的檢體銷毀。您 也可以聯繫本院研究倫理委員會(電話:(02)2312-3456 轉 63155),以協助您解決檢體在 研究使用上的任何爭議。

(2) 剩餘檢體(含其衍生物)之保存與再利用

您的生物檢體將會以專屬號碼進行編碼並在檢體保管者的控管下將保存於 國家衛 生研究院癌症研究所常慧如醫師實驗室, 最長將保存10年.

所有新的研究計畫都要再經由台大醫院研究倫理委員會審議通過,研究倫理委員會若 認定新的研究超出您同意的範圍,將要求我們重新得到您的同意。

是否同意剩餘檢體提供未來巨噬細胞與癌細胞融合在腫瘤纖維化研究之用,並授權台 大醫院研究倫理委員會審議是否需要再取得您的同意

- □ 1.不同意保存我的剩餘檢體,試驗結束後請銷毀
- □ 2.同意以非去連結之方式保存我的剩餘檢體,逾越原同意使用範圍時,需再次得到我 的同意才可使用我的檢體進行新的研究.
- (3) 剩餘檢體未來使用之相關資訊
  - i. 剩餘檢體提供、讓與或授權國內或國外之下列人員使用:
    - ■獲得主持人授權之國內學術研究機構研究人員。
    - ■目前仍不確定您的檢體是否有可能提供給院外及國外的研究者保管或使用 如有此種情形,將由本院研究倫理委員會審查檢體使用的適當性,以保障您的權益。
- ii. 剩餘檢體預期利益或預期研究成果:

由於目前還不知道您的剩餘檢體將用於何種醫學研究,因此無法預測可能的研究成 果。保存剩餘檢體通常不會對您個人有直接的醫療利益,也不會獲得報酬,但是您所 提供檢體,可能促進醫學進步,造福人類健康。

iii. 剩餘檢體研究與個人疾病相關的檢驗檢查結果

當您的剩餘檢體將來使用於某個研究時,我們將不會通知您研究結果或檢體的檢測結 果。一般而言,研究所做的檢測分析,大多還不能運用於醫療照護;但若研究人員認 為研究分析的結果,有助於您的醫療照護,也可能會通知您,並協助安排相關檢測與 專業諮詢。

2. 資料之保存、使用與再利用

在試驗/研究期間,依據計畫類型與您所授權的內容,我們將會蒐集與您有關的病歷資 料、醫療紀錄等資料與資訊,並以一個編號來代替您的名字及相關個人資料。前述資料 若為紙本型式,將會與本同意書分開存放於研究機構之上鎖櫃中;若為電子方式儲存或

版本/日期: 20220225 version 2

NTUHREC Version: AF- 046/09.0

西元 2017 年 06 月 19 日病歷委員會修正通過 MR19-304 西元 2017年 05月 31日品質暨病人安全委員會審核通過

01010-4-601566 文件編號



日:西元

## 國立臺灣大學醫學院附設醫院 National Taiwan University Hospital

臨床試驗/研究受試者說明暨同意書

年月日 研究倫理委員會案號: 202201057RINA

請詳細閱讀內容,待主持人或其授權人員向您說明後,再簽署同意書

建檔以供統計與分析之用,將會存放於設有密碼與適當防毒軟體之專屬電腦內。這些研 究資料與資訊將會保存\_10\_年。上述資料與資訊若傳輸至國外分析與統計,您仍會獲得 與本國法規相符之保障,計畫主持人與相關團隊將盡力確保您的個人資料獲得妥善保

試驗結束後,我們可能將試驗資料用於未來醫學研究,發展其他藥物,診斷性檢測.

#### 3. 基因檢測結果

您提供的血球細胞, 將於實驗室中分化為巨噬細胞, 與實驗室中的癌細胞株進行 融合, 並進行一系列研究, 包括基因檢測, 因基因檢測結果尚屬研究階段, 不確定性過高 /或研究發現不具醫療實用價值,故不會告知您檢測結果。

4. 與個人疾病相關的檢驗檢查結果

因研究結果尚屬研究階段,不確定性過高/或研究發現不具醫療實用價值,因此我們 不會告知您相關的研究檢驗檢查結果。

## (十三)受試者權益:

- 1. 如果您在試驗/研究過程中對研究工作性質產生疑問,對身為患者之權利有意見或懷 疑因參與研究而受害時,可與研究倫理委員會聯絡請求諮詢,電話號碼為: (02)2312-3456轉63155。
- 2. 研究過程中,與您的健康或是疾病有關,可能影響您繼續接受臨床研究意願的任何重 大發現,都將即時提供給您。如果您決定退出,醫師會安排您繼續接受醫療照護。如 果您決定繼續參加試驗/研究,可能需要簽署一份更新版的同意書。
- 3. 本同意書一式2份,試驗主持人或其授權人員已將1份已簽名的同意書交給您,並已完 整說明本研究之性質與目的。 醫師已回答您有關研究的問題。
- 4. 參加試驗研究計畫之補助:本研究未提供補助。
- 若試驗結束後 1 年內,發現有非預期且直接影響您的安全疑慮,亦將通知您。

#### (十四)本研究預期可能衍生之商業利益及其應用之約定:

若您提供周邊血液, 本研究將抽取單核血球, 分化為巨噬細胞進行研究. 該巨噬細胞可 能會與癌細胞株共同培養,產生融合細胞株,該細胞株可能短暫繁殖一段時間,少數機會可 能永久不斷繁殖. 本計畫將利用上述融合細胞株, 與一般癌細胞株比較, 進行研究, 可能導 致發現、發明或研發商業產品。您與您的家人不會因這些資訊中的研發成果、發明或其他發 現而獲得任何財務利益或金錢補償,或擁有上述發明結果的所有權。上述融合細胞株,若能 永久不斷繁殖,也將保存不超過10年.

版本/日期: 20220225 version 2

NTUHREC Version: AF-046/09.0

西元 2017 年 06 月 19 日病歷委員會修正通過 MR19-304 西元 2017年 05月 31日品質暨病人安全委員會審核通過

01010-4-601566 文件編號

國立臺灣大學醫學院附設醫院 National Taiwan University Hospital

姓名: 生日:西元 年月日

臨床試驗/研究受試者說明暨同意書

研究倫理委員會案號: 202201057RINA

請詳細閱讀內容,待主持人或其授權人員向您說明後,再簽署同意書 第7頁

| (十五)簽名: | |
|---|---|
| <ol> <li>試驗主持人、或協同主持人或其授權人員已詳細解釋<br/>的性質與目的,及可能產生的危險與利益。</li> </ol> | 有關本研究計畫中上述研究方法 |
| 試驗主持人/協同主持人簽名: | |
| 日期:年月日 | |
| 在取得同意過程中其他參與解說及討論之研究人員 | 簽名: |
| 日期:年月日 | |
| <ol> <li>經由說明後本人已詳細瞭解上述研究方法及可能產<br/>究計畫的疑問,亦獲得詳細解釋。本人同意接受並自<br/>的同意書。</li> </ol> | |
| 受試者簽名: 日期: | 年月日 |
| 出生年月日:年月日 電話: | |
| 國民身分證統一編號: 性別: | |
| 通訊地址: | |
| 法定代理人/有同意權之人簽名: 日期 | :年月日 |
| 與受試者關係(請圈選):配偶、父、母、兒、女、 | 其他: |
| 出生年月日:年月日 電話: | |
| 國民身分證統一編號: | |
| 通訊地址: | |
| *適用醫療法第79條第1項但書或人體研究法第12條第1項但<br>法第79條第2項、人體試驗管理辦法第5條或人體研究法第<br>*受試者為無行為能力者(未滿七歲之未成年人者或受監護宣告之<br>之人,由監護人擔任其法定代理人。<br>* 受試者為限制行為能力者(滿七歲以上之未成年人或因精神障<br>受意思表示、辨識其意思表示效果之能力,顯有不足,而受 | 12條第3、4項規定辦理:<br>之人),由法定代理人簽名;受監護宣告<br>礙、其他心智缺陷,致其為意思表示、 |
| 交息心表小、辨識兵息心表小效米之能力,顯有不足,而受為<br>代理人或輔助人之同意。<br>*受試者雖非無行為能力或限制行為能力者,但因 <b>意識混亂或有</b> | |
| 和判斷時,由有同意權之人簽名。有同意權人順序如下:<br>1.屬新藥、新醫療器材、新醫療技術之人體試驗(人體試驗管 | |

版本/日期: 20220225 version 2

NTUHREC\_Version: AF- 046/09.0

西元 2017 年 06 月 19 日病歷委員會修正通過 MR19-304 西元 2017 年 05 月 31 日品質暨病人安全委員會審核通過

文件編號 01010-4-601566

(1)配偶。(2) 父母。(3) 同居之成年子女。(4)與受試者同居之祖父母。(5)與受試者同居之兄弟姊

版次

04

日:西元

### 國立臺灣大學醫學院附設醫院 National Taiwan University Hospital

National Taiwan University Hospital 臨床試驗/研究受試者說明暨同意書

研究倫理委員會案號: 202201057RINA

日

年 月

請詳細閱讀內容,待主持人或其授權人員向您說明後,再簽署同意書

第8頁

妹。(6) 最近一年有同居事實之其他親屬。

- 2. 屬人體研究(人體研究法第12條):
- (1)配偶。(2)成年子女。(3)父母。(4)兄弟姊妹。(5)祖父母。

依前項關係人所為之書面同意,其書面同意,得以一人行之;關係人意思表示不一致時,依前項各款先後定其順序。前項同一順序之人,以親等近者為先,親等同者,以同居親屬為先,無同居親屬者,以年長者為先。

| 見證人簽名: | 日期: | :年 | ·月_ | B |
|--------|-----|----|-----|---|
|--------|-----|----|-----|---|

- \* 受試者、法定代理人或有同意權之人皆無法閱讀時,應由見證人在場參與所有有關受試者同意之討論。並確定受試者、法定代理人或有同意權之人之同意完全出於其自由意願後,應於受試者同意書簽名並載明日期。試驗/研究相關人員不得為見證人。
- \* 若意識清楚,但無法親自簽具者,得以按指印代替簽名,惟應有見證人。

版本/日期: 20220225 version 2 NTUHREC Version: AF- 046/09.0